CLINICAL TRIAL: NCT04114721
Title: Learning Curve of Video-laryngoscope (VL) for First Attempt Successful Endotracheal Intubation During Cardiopulmonary Resuscitation (CPR)
Brief Title: Learning Curve of VL for Intubation During CPR
Status: Completed | Type: Observational
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Sang O, Park, Associate Professor, Konkuk University Medical Center
Other Study IDs: CPRintuexperience_VL
Record Dates: First submitted 2019-10-02; First posted 2019-10-03 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Cardiopulmonary Arrest
Keywords: intubation; cardiopulmonary resuscitation; Learning curve; videolaryngoscope
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a clinical study based on analysis of video-clip data of endotracheal intubation (ETI) using videolaryngoscope (VL) and clinical data for cardiopulmonary resuscitation patients between 2012.03.01.-2015.02.28.

The purpose of this study is to evaluate the appropriate numbers of VL usages for successful ETI at first attempt during cardiopulmonary resuscitation.

DETAILED DESCRIPTION:
Direct layngoscope (DL) is a basic tool for endotracheal intubation(ETI) during cardiopulmonary resuscitation(CPR). ETI during CPR has higher risks of failure or delayed success with frequent attempts, misplacement of the tube, and prolonged interruptions of chest compressions. The main problems associated with ETI relate to the inherently technical difficulty in using DL. VL have various advantages of fast learning curve and overall success comparing with the DL in non-arrest patients, but there was no known data of learnig curve of successful ETI during CPR.

This study tried to estimate the the appropriate numbers of VL usage for successful ETI at first attempt during CPR. So the investigators analyze the success rate, speed, trial number, incidence of complications, and hands-off time of ETI using VL which in real clinical setting. In addition, this study analyze the residency training term, total number of of VL usage using VL at that time.

ELIGIBILITY:
Inclusion Criteria:

* patients who suffer sudden cardiac arrest and physician tried ti intubate using viseolaryngoscope.

Exclusion Criteria:

* case of requesting the do-not-attempt resuscitation befor ETI
* intubated cases before arrival to emergency department
* physician tried ti intubate using direct-laryngoscope

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: emergency physicians in an urban ED at a tertiary training hospital in Seoul, Republic of Korea
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
YES or No of successful intubation without complication | successful endotracheal intubation with in 60 seconds
  endotracheal intubation, hands-off time < 10 seconds, first trial

CONTACTS AND LOCATIONS:
Overall Officials: Sang O Park, M.D., PhD, Principal Investigator — Department of Emergency Medicine, Konkuk University Medical center
Locations (1):
- Department of Emergency Medicine, Konkuk University Medical center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dagli R, Canturk M, Celik F, Erbesler ZA, Gurler M. [The role of videolaryngoscope in endotracheal intubation training programs]. Braz J Anesthesiol. 2018 Sep-Oct;68(5):447-454. doi: 10.1016/j.bjan.2018.02.008. Epub 2018 Jul 17. PMID 30025947
- [Background] Bernhard M, Benger JR. Airway management during cardiopulmonary resuscitation. Curr Opin Crit Care. 2015 Jun;21(3):183-7. doi: 10.1097/MCC.0000000000000201. PMID 25922892
- [Background] Buis ML, Maissan IM, Hoeks SE, Klimek M, Stolker RJ. Defining the learning curve for endotracheal intubation using direct laryngoscopy: A systematic review. Resuscitation. 2016 Feb;99:63-71. doi: 10.1016/j.resuscitation.2015.11.005. Epub 2015 Dec 19. PMID 26711127
- [Result] Park SO, Baek KJ, Hong DY, Kim SC, Lee KR. Feasibility of the video-laryngoscope (GlideScope(R)) for endotracheal intubation during uninterrupted chest compressions in actual advanced life support: a clinical observational study in an urban emergency department. Resuscitation. 2013 Sep;84(9):1233-7. doi: 10.1016/j.resuscitation.2013.03.026. Epub 2013 Mar 26. PMID 23541527